CLINICAL TRIAL: NCT06830447
Title: Test-retest Reliability of Low-frequency Fatigue Assessed Using Myocene
Brief Title: Test-retest Reliability of Myocene
Status: Not yet recruiting | Type: Observational
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Filipe Silvano Pinto Maia, Principal Investigator, University of Maia
Other Study IDs: Myo_testretest
Record Dates: First submitted 2025-02-05; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Reliability; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single group: participants will perform the myocene measurement twice
  Interventions: Other: low-frequency fatigue

INTERVENTIONS:
Other: low-frequency fatigue — Low frequency fatigue tested with myocene

SUMMARY:
The test retest reliability of Myocene will be tested.

ELIGIBILITY:
Inclusion Criteria:

* active individuals

Exclusion Criteria:

* injured participants
* unhealthy volunteers

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be sports science students, physically active.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
low-frequency fatigue | baseline and 30 minutes post baseline.
  Low frequency fatigue will be assessed using myocene. Participants will seat on the device with their leg positioned against the "Myo-sensor". Electrical muscle stimulation will be applied using biphasic square waves with a pulse width of 400 µs, delivered through three electrodes. A pre-programmed Myocene protocol, which has a duration of about 2 minutes will be applied

IPD SHARING:
Plan to Share IPD: Undecided